CLINICAL TRIAL: NCT02830880
Title: Investigation of Therapy Response With Amino Acid Analogue Transport PET Imaging
Brief Title: FACBC Prostate Therapy Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Blue Earth Diagnostics (Industry); Nihon Medi-Physics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, David M. Schuster, MD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00073616
Record Dates: First submitted 2016-06-30; First posted 2016-07-13 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: Imaging; Nuclear medicine; Oncology; Radiology; Urogenital disorders
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Urogenital Diseases | interventions — fluciclovine F-18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FACBC (Experimental): Participants with biopsy-proven primary or recurrent castration-resistant prostate carcinoma with skeletal and/or nodal involvement will undergo an FACBC PET-CT scan.
  Interventions: Drug: FACBC PET-CT; Other: MRI, CT, or Bone Scan

INTERVENTIONS:
Drug: FACBC PET-CT — Anti-3-[18F]FACBC is an investigational positron emission tomography (PET) radiotracer being studied given intravenously prior to PET scan.
  Other Names: Fluciclovine
Other: MRI, CT, or Bone Scan — Conventional imaging such as a MRI, CT, or bone scan will be performed to correlate imaging findings.

SUMMARY:
The purpose of this study is to assess if using anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (FACBC or fluciclovine) PET scan will be useful in determining if participants are responding to chemotherapy treatment. Investigators will enroll participants whose cancer has been treated with hormone therapy and now the cancer is not responding to the treatment (castration -resistant), and so therefore will be started on chemotherapy. Investigators aim to enroll thirty participants in this study.

DETAILED DESCRIPTION:
The goal of the investigation is to examine therapeutic monitoring of chemotherapy in castrate resistant prostate carcinoma with anti-3-[18F]FACBC in prostate carcinoma to determine if anti-3-[18F]FACBC amino acid imaging can serve as an accurate and efficient imaging biomarker.

Investigators will perform a baseline anti-3-[18F]FACBC PET-CT of the whole body. All participants will also undergo conventional staging including 99mTc methylene diphosphonate (MDP) bone scanning and computed tomography scan (CT) or magnetic resonance imaging (MR) of the abdomen and pelvis which are standard of care at the enrolling institution. This study will not interfere with standard patient evaluation or delay therapy.

All 30 participants will receive chemotherapy every 3 weeks for 6 cycles. Participants will undergo a repeat anti-3-[18F]FACBC PET-CT after 1 and 6 cycles and also repeat conventional imaging including bone scanning CT or MR of the abdomen and pelvis after 6 cycles. At the end of the study, the study team will then record the response (or lack thereof) on anti-3-[18F]FACBC PET-CT and correlate that response with response per standard clinical criteria including bone scan uptake for skeletal lesions, CT or MR for soft tissue and skeletal lesions, prostate-specific antigen (PSA) progression or regression, and other clinical parameters such as declining performance status.

ELIGIBILITY:
Inclusion Criteria:

* Primary or recurrent castration resistant prostate carcinoma with skeletal and/or nodal involvement not currently undergoing systemic chemotherapy who are about to commence therapy with docetaxel/prednisone. (Note that systemic hormonal targeted therapy including luteinizing hormone-releasing hormone (LHRH) agonists (Lupron or Trelstar), other anti-androgens, and/or Abiraterone or Enzalutamide may be in use.)
* Ability to lie still for PET scanning
* Ability to provide written informed consent

Exclusion Criteria:

* Age less than 18 years
* Inability to lie still for PET scanning
* Inability provide written informed consent
* Currently undergoing chemotherapy for organ confined or systemic disease. This does not preclude patients who had previously received upfront docetaxel in the hormone sensitive setting.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schuster DM, Nieh PT, Jani AB, Amzat R, Bowman FD, Halkar RK, Master VA, Nye JA, Odewole OA, Osunkoya AO, Savir-Baruch B, Alaei-Taleghani P, Goodman MM. Anti-3-[(18)F]FACBC positron emission tomography-computerized tomography and (111)In-capromab pendetide single photon emission computerized tomography-computerized tomography for recurrent prostate carcinoma: results of a prospective clinical trial. J Urol. 2014 May;191(5):1446-53. doi: 10.1016/j.juro.2013.10.065. Epub 2013 Oct 19. PMID 24144687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from patients receiving services at Emory University Hospital in Atlanta, Georgia. Participant enrollment began in July 2016, follow up for the primary outcome measures was complete by December 1, 2018 and follow up for the secondary outcome measure was completed on September 30, 2019.
Groups:
- FACBC PET-CT: Participants with biopsy-proven primary or recurrent castration-resistant prostate carcinoma with skeletal and/or nodal involvement receiving anti-1-amino-3-[18F]fluorocyclobutane-1-carboxylic acid (FACBC) radiotracer intravenously prior to positron emission tomography (PET) scan.
Period: Overall Study
Arm/Group | FACBC PET-CT
Started | 7
Completed Visit After Cyle 1 | 7
Completed (Completed visit after Cycle 6) | 4
Not Completed | 3
Not completed — Adverse reaction to chemotherapy | 1
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- FACBC PET-CT: Participants with biopsy-proven primary or recurrent castration-resistant prostate carcinoma with skeletal and/or nodal involvement receiving Anti-3-[18F]FACBC radiotracer intravenously prior to PET scan.
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percent Change Assessed by FACBC PET Scan
Description: Clinical response will be assessed with FACBC PET imaging. The same measurements of the lesions and background structures will be undertaken at baseline and post-therapy scan. The researchers utilized the following parameters to follow response to therapy: maximum standardized uptake value (SUVmax) of most intense lesion each of bone and node, sum and mean SUVmax of up to 5 index lesions for each of bone and node of most intense lesion each of bone and node of the 5 index lesions for each of bone and node. SUVmax measures uptake of the radiotracer by malignant cells. Percent change after therapy, compared to baseline, was calculated and a positive percent increase indicates greater uptake of FACBC by cancer cells.
Time Frame: Baseline, Cycle 1 (Week 2), Cycle 6 (Week 17)
Population: This analysis includes participants completing the study visits used in each change from baseline determination.
Measure: Mean (Standard Deviation); unit: percent change of SUVmax
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 7
percent change of SUVmax
  Percent change between Baseline and Cycle 1 | 3.2 (32.6)
  Percent change between Baseline and Cycle 6: number analyzed (Participants) | 4
  Percent change between Baseline and Cycle 6 | 23.5 (21.4)

2. Primary Outcome: Prostate Specific Antigen Level
Description: Prostate Specific Antigen (PSA) serum biomarker will be used to assess response to treatment. PSA level will be collected via blood draw. While a formal cutpoint signifying prostate cancer is not generally used as PSA levels vary between men, in general, higher PSA levels indicate prostate cancer.
Time Frame: Baseline, Cycle 1 (Week 2), Cycle 6 (Week 17)
Population: This analysis includes participants completing the study visits.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 7
nanograms per milliliter (ng/mL)
  Baseline | 249.8 (471.9)
  After completing Cycle 1 | 245.3 (472.5)
  After completing Cycle 6: number analyzed (Participants) | 4
  After completing Cycle 6 | 39.9 (23.7)

3. Primary Outcome: Number of Participants Responding to Treatment Assessed by MRI
Description: Participants will have an MRI or a CT scan to assess response to treatment. Treatment response will be reported as follows:
  * Complete Response (CR) Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Complete Response Unknown (CRU)
  * Partial Response (PR) At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
  * Stable Disease (NR/SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  * Progressive Disease (PD) At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Baseline, Cycle 1 (Week 2), Cycle 6 (Week 17)
Population: Data were not collected for this outcome measure as all participants had a CT scan rather than an MRI to assess response to treatment.
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Participants Responding to Treatment Assessed by CT Scan
Description: A CT will be used to assess response to treatment. Treatment response will be reported as follows:
  * Complete Response (CR) Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR) At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
  * Stable Disease (NR/SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  * Progressive Disease (PD) At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: After Cycle 6 (Week 17)
Population: This analysis includes participants completing the study.
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 4
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 4
  Progressive Disease | 0

5. Primary Outcome: Number of Participants With a Clinical Response Assessed by Bone Scan
Description: Each patient underwent 99mTc MDP whole body bone scanning at baseline, and after the 6th cycle. Bone scans findings were interpreted based on recommendations from Prostate Cancer Clinical Trial Working Group 3 (PCCTWG3) using a specialized Bone Scan Assessment Tool. The change in disease response after cycle 6 compared to the baseline assessment is presented here.
Time Frame: Baseline, After Cycle 6 (Week 17)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 4
Participants
  Difference in disease response: None | 0
  Difference in disease response: Response | 0
  Difference in disease response: Stable | 2
  Difference in disease response: Progressive | 2

6. Secondary Outcome: Number of Deaths
Description: The number of deaths that have occurred was assessed at the end of study.
Time Frame: End of Study (up to 1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | FACBC PET-CT
Number analyzed (Participants) | 7
Participants | 3

ADVERSE EVENTS:
Time Frame: Information about adverse events that were potentially related to the radiotracer used for FACBC PET-CT scan was collected from the time of giving consent to participate in the study through the post-cycle 6 visit, approximately 17 weeks.
Arm/Group | FACBC PET-CT
All-Cause Mortality (participants affected / at risk) | 3/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT02830880/Prot_SAP_000.pdf